CLINICAL TRIAL: NCT02550808
Title: Metabolic and Histological Changes in Skeletal Muscle and Fat Tissue in Patients With Chronic Cardiopulmonary Disease
Brief Title: Metabolic Changes in Patients With Chronic Cardiopulmonary Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General and Teaching Hospital Celje (Other)
Collaborators: University of Ljubljana (Other); General Hospital Murska Sobota (Other); Maastricht University (Other)
Responsible Party: Principal Investigator, Mitja Lainscak, Professor of Internal Medicine, General and Teaching Hospital Celje
Other Study IDs: ML-MTB-001
Record Dates: First submitted 2015-09-03; First posted 2015-09-16 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Heart Failure; Chronic Obstructive Pulmonary Disease; Malignancy; Chronic Kidney Disease
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive; Neoplasms; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum; plasma; Skeletal muscle; fat tissue; urine; full blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Heart failure
- Chronic obstructive pulmonary disease
- Chronic kidney disease
- Malignancy
- Controls

SUMMARY:
This study aims to evaluate prevalence of sarcopenia and cachexia in patients with chronic cardiopulmonary disease. The investigators will also investigate metabolic disorders like glucose metabolism, presence of metabolic syndrome, body composition and histological changes in skeletal muscle and body fat. Finally, patients will be followed for clinical endpoints.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic disease (Heart failure, COPD, malignancy, CKD) or no diagnosis (controls)

Exclusion Criteria:

* refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic disease (Heart failure, COPD, malignancy, CKD) and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2012-03; Primary Completion 2016-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Insulin resistance (HOMA-IR) | Baseline
  HOMA-IR as calculated by formula using insulin and blood glucose

SECONDARY OUTCOMES:
Muscle strength (Handgrip test) | Baseline
  Handgrip test
Change in exercise capacity (6 minute walk test) | baseline and after 5 weeks
  Determined by incremental exercise test, 6 minute walk test
Neurohormonal activation (NT-proBNP concentration) | Baseline
  NT-proBNP concentration
Change in apoptosis in skeletal muscle (number of apoptotic cells per square mm) | Baseline and after 5 weeks
  histological evaluation: number of apoptotic cells per square mm
Change in insulin resistance (HOMA-IR) | Baseline and after 5 weeks
  HOMA-IR as calculated by formula using insulin and blood glucose

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital Celje, Celje, Slovenia